CLINICAL TRIAL: NCT02630394
Title: A Pilot Study of Azithromycin Prophylaxis for Acute Chest Syndrome in Sickle Cell Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator has moved to another institution
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Suvankar Majumdar, Associate Professor of Pediatrics, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SCD_ACS_AZM
Record Dates: First submitted 2015-11-26; First posted 2015-12-15 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Sickle Cell Disease; Acute Chest Syndrome
Keywords: sickle cell disease; acute chest syndrome
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azithromycin prophylaxis (Experimental): Azithromycin will be supplied as a 250-mg tablet. Participants weighing less than 40 mg will be instructed to take 1 tablet 3 days a week (Monday, Wednesday, and Friday), and participants who weigh more than 40 kg will be instructed to take 2 tablets on the same 3 days per week.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin
  Other Names: Zithromax

SUMMARY:
Acute chest syndrome (ACS), a lung complication in sickle cell disease (SCD), is the second most common cause of hospitalization and leading cause of death in SCD. ACS is associated with airway inflammation, and a major cause is pulmonary infection from atypical organisms. To date, there are no drugs available to reduce inflammation and risk of recurrent ACS. Macrolides are a group of antibiotics that exert immunomodulatory and anti-inflammatory actions both in vitro and in vivo. In addition, macrolides reduce bacterial burden in the airway of atypical organisms, all of which play an important role in the pathophysiology of ACS. Numerous studies have evaluated macrolide prophylaxis in conditions associated with lung inflammation, such as cystic fibrosis, asthma, bronchiectasis etc., and high quality evidence have found macrolides to be beneficial as a disease modifying agent that leads to improvement in airway inflammation, reduced pulmonary exacerbations and improved lung function. The investigators hypothesize that azithromycin prophylaxis is well tolerated and has the potential to reduce inflammation and improve lung outcome in children with SCD with a history of ACS. A prospective, single arm, open label feasibility study of azithromycin prophylaxis will be performed in children with SCD with a history ACS with the specific aim to examine the feasibility, safety and tolerability of azithromycin prophylaxis administration in participants with SCD , and to examine whether azithromycin prophylaxis has the potential to improve lung outcome. In addition, this study will determine whether azithromycin prophylaxis reduces inflammation in participants with SCD with a history of ACS.

DETAILED DESCRIPTION:
Specific Aims:

Acute chest syndrome (ACS), a lung complication in sickle cell disease (SCD), is the second most common cause of hospitalization and leading cause of death in SCD. Recurrent ACS has been associated with poor lung function outcome that is comparable to cystic fibrosis. ACS is associated with airway inflammation, and a major cause is pulmonary infection from atypical organisms. To date, there are no drugs available to reduce inflammation and risk of recurrent ACS. Thus newer therapies are urgently needed to address this important issue associated with increased morbidity from debilitating chronic lung disease and mortality in SCD. Macrolides are a group of antibiotics that exert immunomodulatory and anti-inflammatory actions both in vitro and in vivo. It has been shown to inhibit neutrophil activation and mobilization, modulate oxidant production by neutrophils and of proinflammatory cytokine synthesis and release by leukocytes, reduce systemic markers of inflammation, inhibit intercellular adhesion molecules on epithelial cell surfaces, and block the activation of certain nuclear transcription factors. In addition, macrolides reduce bacterial burden in the airway of atypical organisms, all of which play an important role in the pathophysiology of ACS. Indeed, numerous studies have evaluated macrolide prophylaxis in conditions associated with lung inflammation, such as cystic fibrosis, asthma, bronchiectasis etc., and high quality evidence have found macrolides to be beneficial as a disease modifying agent that leads to improvement in airway inflammation, reduced pulmonary exacerbations and improved lung function. However, azithromycin has never been studied before in SCD. The investigators hypothesize that azithromycin prophylaxis is well tolerated and has the potential to reduce inflammation and improve lung outcome in children with SCD with a history of ACS.

A prospective, single arm, open label feasibility study of azithromycin prophylaxis will be performed in children with SCD with a history ACS with the following specific aims:

Specific Aim 1: Examine the feasibility, safety and tolerability of azithromycin prophylaxis administration in children with SCD. A cohort of 15 participants with sickle cell disease 6 to 16 years old will be placed on azithromycin prophylaxis, and followed closely to evaluate medication adherence and for any adverse effects from taking the medication.

Specific Aim 2: Examine whether azithromycin prophylaxis has the potential to improve lung outcome in participants with SCD with a history of ACS. In the same cohort of 15 patients, baseline pulmonary function testing will be performed evaluating Forced expiratory volume 1 sec (FEV1) and Forced vital capacity (FVC) measurements prior to starting azithromycin prophylaxis, and then again at study end period after 1 year to evaluate for any change.

Specific Aim 3: Determine whether azithromycin prophylaxis reduces inflammation in participants with SCD with a history of ACS. In the same cohort of 15 participants, baseline markers of inflammation will be performed, specifically C-reactive protein (CRP), Tumor necrosis factor Alpha (TNF-α), interleukin IL-1, IL-1β, IL-4, IL-6, and IL-8, and then repeated at specific time intervals of 16 weeks, 32 weeks and 48 weeks (study end).

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of SCD (Hemoglobin SS, hemoglobin Sβ0 thalassemia)
* History of acute chest syndrome - the history of acute chest syndrome will be confirmed by a retrospective medical chart review that meets the standard definition as mentioned in the Background section.
* Age ≥ 6 years to 16 years old

Exclusion Criteria:

* Hemoglobin Sβ+thalassemia and hemoglobin SC subject will be excluded as this group of patients do not typically have severe SCD that places them at risk of developing recurrent acute chest syndrome
* No history of acute chest syndrome
* Significant neurologic impairment as judged by health care provider.
* Inability to take/swallow a tablet
* History of poor adherence to clinic visits.
* History of renal or hepatic dysfunction
* Chronic red blood cell transfusion
* History of allergy to azithromycin or macrolide antibiotic
* History of cardiac arrhythmia
* History of prolonged QT

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 48 weeks

SECONDARY OUTCOMES:
Percent adherence with azithromycin prophylaxis | 48 weeks
Number of participants with improved forced vital capacity (cm3) | 48 weeks
Number of participants with improved forced expiratory volume 1 (cm3/sec) | 48 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Background] Castro O, Brambilla DJ, Thorington B, Reindorf CA, Scott RB, Gillette P, Vera JC, Levy PS. The acute chest syndrome in sickle cell disease: incidence and risk factors. The Cooperative Study of Sickle Cell Disease. Blood. 1994 Jul 15;84(2):643-9. PMID 7517723
- [Background] Vichinsky EP, Neumayr LD, Earles AN, Williams R, Lennette ET, Dean D, Nickerson B, Orringer E, McKie V, Bellevue R, Daeschner C, Manci EA. Causes and outcomes of the acute chest syndrome in sickle cell disease. National Acute Chest Syndrome Study Group. N Engl J Med. 2000 Jun 22;342(25):1855-65. doi: 10.1056/NEJM200006223422502. PMID 10861320
- [Background] Dean D, Neumayr L, Kelly DM, Ballas SK, Kleman K, Robertson S, Iyer RV, Ware RE, Koshy M, Rackoff WR, Pegelow CH, Waldron P, Benjamin L, Vichinsky E; Acute Chest Syndrome Study Group. Chlamydia pneumoniae and acute chest syndrome in patients with sickle cell disease. J Pediatr Hematol Oncol. 2003 Jan;25(1):46-55. doi: 10.1097/00043426-200301000-00010. PMID 12544773
- [Background] Boyd JH, Macklin EA, Strunk RC, DeBaun MR. Asthma is associated with acute chest syndrome and pain in children with sickle cell anemia. Blood. 2006 Nov 1;108(9):2923-7. doi: 10.1182/blood-2006-01-011072. Epub 2006 May 11. PMID 16690969
- [Background] Knight-Madden JM, Forrester TS, Lewis NA, Greenough A. Asthma in children with sickle cell disease and its association with acute chest syndrome. Thorax. 2005 Mar;60(3):206-10. doi: 10.1136/thx.2004.029165. PMID 15741436
- [Background] Vance LD, Rodeghier M, Cohen RT, Rosen CL, Kirkham FJ, Strunk RC, DeBaun MR. Increased risk of severe vaso-occlusive episodes after initial acute chest syndrome in children with sickle cell anemia less than 4 years old: Sleep and asthma cohort. Am J Hematol. 2015 May;90(5):371-5. doi: 10.1002/ajh.23959. Epub 2015 Mar 30. PMID 25619382
- [Background] Zarogoulidis P, Papanas N, Kioumis I, Chatzaki E, Maltezos E, Zarogoulidis K. Macrolides: from in vitro anti-inflammatory and immunomodulatory properties to clinical practice in respiratory diseases. Eur J Clin Pharmacol. 2012 May;68(5):479-503. doi: 10.1007/s00228-011-1161-x. Epub 2011 Nov 22. PMID 22105373
- [Background] Saiman L, Marshall BC, Mayer-Hamblett N, Burns JL, Quittner AL, Cibene DA, Coquillette S, Fieberg AY, Accurso FJ, Campbell PW 3rd; Macrolide Study Group. Azithromycin in patients with cystic fibrosis chronically infected with Pseudomonas aeruginosa: a randomized controlled trial. JAMA. 2003 Oct 1;290(13):1749-56. doi: 10.1001/jama.290.13.1749. PMID 14519709
- [Background] Ratjen F, Saiman L, Mayer-Hamblett N, Lands LC, Kloster M, Thompson V, Emmett P, Marshall B, Accurso F, Sagel S, Anstead M. Effect of azithromycin on systemic markers of inflammation in patients with cystic fibrosis uninfected with Pseudomonas aeruginosa. Chest. 2012 Nov;142(5):1259-1266. doi: 10.1378/chest.12-0628. PMID 22595153